CLINICAL TRIAL: NCT00956072
Title: A Phase III Randomized Study Evaluating Surgery of Residual Disease in Patients With Metastatic Gastro-intestinal Stromal Tumor Responding to Imatinib Mesylate.
Brief Title: Imatinib Mesylate With or Without Surgery in Treating Patients With Metastatic Gastrointestinal Stromal Tumor That is Responding to Imatinib Mesylate
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-62063; EORTC-62063; EU-20955; EUDRACT-2007-002257-23; NOVARTIS-EORTC-62063
Record Dates: First submitted 2009-08-08; First posted 2009-08-11 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: gastrointestinal stromal tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

ARMS (2):
- Arm I (Experimental): Patients undergo surgery of residual disease.
  Interventions: Procedure: therapeutic conventional surgery
- Arm II (Active Comparator): Patients receive imatinib mesylate therapy according to standard of care.
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate — Patients receive imatinib mesylate
  Arms: Arm II
Procedure: therapeutic conventional surgery — Patients undergo surgery
  Arms: Arm I

SUMMARY:
RATIONALE: Surgery may remove residual disease in patients with gastrointestinal stromal tumor that is responding to imatinib mesylate. It is not yet known whether surgery is more effective than continued imatinib mesylate in treating patients with metastatic gastrointestinal stromal tumor.

PURPOSE: This randomized phase III trial is studying giving imatinib mesylate therapy together with surgery to see how well it works compared with imatinib mesylate alone in treating patients with metastatic gastrointestinal stromal tumor that is responding to imatinib mesylate.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate whether surgery of residual disease improves the progression-free survival of patients with metastatic gastrointestinal stromal tumor responding to imatinib mesylate.

Secondary

* Correlate the pharmacokinetics of imatinib mesylate and its metabolites before and after randomization.

OUTLINE: This is a multicenter study. Patients are stratified according to center, site of tumor origin (stomach vs small bowel vs others), and site of metastases (liver vs abdominal cavity vs both). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo surgery of residual disease. Patients will then resume imatinib mesylate therapy according to standard of care as soon as possible after surgery (as soon as the patient restarts taking oral feeding).
* Arm II: Patients receive imatinib mesylate therapy according to standard of care.

Patients complete quality of life questionnaires at baseline; immediately after hospital discharge (arm I only); and at 5, 11, and 23 months. Blood samples may be collected for pharmacokinetic studies.

After completion of study therapy, patients are followed up every 3 months for 5 years and then every 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gastrointestinal stromal tumor expressing CD117+ or with documented mutation of the KIT or PDGFRA gene
* Metastatic disease (liver and/or abdominal cavity)

  * No extra-abdominal metastases
* Measurable disease according to RECIST criteria
* Achieved complete response, partial response, or stable disease without progression since the start of imatinib mesylate therapy, documented according to RECIST
* Underwent 6-12 months of treatment with imatinib mesylate as a standard of care or within other clinical studies (surgery should be feasible before the end of the 12th month from imatinib mesylate onset)
* Surgically resectable residual disease as assessed by CT scan and/or MRI within the past 14 days

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* ANC > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Creatinine < 120 μmol/L
* Albumin > 25 g/L
* Total bilirubin < 2 times upper limit of normal (ULN)
* AST and ALT < 2.5 times ULN (< 5 ULN in case of liver metastases)
* Alkaline phosphatase < 2.5 times ULN (< 5 ULN in case of bone or liver metastases)
* Negative pregnancy test within the past 14 days
* Fertile patients must use effective contraception
* No uncontrolled hypertension (diastolic BP > 95 mm Hg and systolic BP > 170 mm Hg)
* No myocardial infarction, unstable, or uncontrolled cardiac disease within the past 6 months
* No history of arterial thrombosis or deep vein thrombosis within the past year
* No bleeding diathesis, coagulopathy, or major bleeding within the past 6 months
* No severe and/or uncontrolled concurrent medical disease, including any of the following conditions:

  * Diabetes
  * Chronic renal disease
  * Liver disease, including chronic viral hepatitis judged at risk of reactivation
  * Active infection, including HIV infection
* No prior malignancy (other than in situ cervical cancer, in situ melanoma, or basal cell or squamous cell cancer of the skin) unless treated with curative intent and without evidence of disease for at least 3 years
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior adjuvant or neo-adjuvant imatinib mesylate or other tyrosine kinase inhibitor
* No coumadin-type anticoagulant > 2mg/day within the past 7 days
* No major surgery within the past 28 days
* No medication that interacts moderately or strongly with the CYP3A system within the past 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-05; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Overall survival
Pathological response to imatinib mesylate according to RECIST criteria
Rate of complete resection
Surgical morbidity
Quality of life as measured by EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Gronchi, Principal Investigator — Istituto Nazionale per lo Studio e la Cura dei Tumori
Locations (1):
- European Organization for Research and Treatment of Cancer, Naples, Italy